CLINICAL TRIAL: NCT03117907
Title: Comparison of Peripheral Perfusion Level Between Two Groups of Newborns According to Their Infectious Status Defined by the Criteria of the Center for Disease Control and Prevention (CDC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI01-2016
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2016-04

CONDITIONS: Newborn; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants with low infectious status
- Infants with high infectious status

SUMMARY:
Despite advances in medicine, secondary neonatal infection remains a continuing concern because of the associated high morbidity and mortality. The usual mechanism of infection responds to the transmission of germs by the equipment used for care (eg, catheters) and by the hands of caregivers. In preterm infants in particular, some infections can also have an endogenous source, by translocation of colonization germs present in the digestive tract.

The first line of prevention of secondary infection corresponds to compliance with the rules of hand hygiene, work surfaces and equipment carried out, the effect of which on the control of the incidence of secondary infection is regularly demonstrated. When declared, bacterial infection should be treated as quickly as possible with appropriate and effective antibiotics to preserve the healing prognosis. Compared to the infant and the larger child, clinical signs of calling are atypical and discrete. In the absence of staff trained to monitor newborns specifically, there is a real risk of discovering the existence of the infection only at an advanced stage corresponding, among other things, to circulatory collapse. This risk is not completely excluded, even with experienced practitioners, because the positive signs are rude and may go unnoticed (eg, signs of calling such as fever are rare in the newborn). Support for early diagnosis of neonatal infection by automatic monitoring systems has reduced mortality by 30% in the units where it has been applied. This is probably due to the fact that early warning made it possible to start the antibiotic treatment earlier and to complete the bacteriological diagnosis in order to better orient the therapeutic attitude. The best criteria for early diagnosis by automated systems were provided by the statistical analysis of cardiac variability, the results of the research and correspond to the standard deviation, the asymmetry and the entropy of the series d Cardiac intervals. Since microbial aggression has an impact on many vegetative variables outside of the electrocardiogram, our current research aims to determine whether the analysis of the perfusion index (PI) Which are of interest for detecting disturbances in the early stages of infection in newborns. IP corresponds to the ratio of the amplitude of the oscillating phase to the intensity of the constant part of the opto-plethysmography wave; It is obtained from signals recorded in a non-invasive manner by the same infrared sensor for pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Newborn of corrected age between 27 SA and 42 SA with at least 72 hours of postnatal age
* Presence of clinical or biological criteria of infection according to CDC definitions
* Absence of clinical or biological criteria for infection according to CDC definitions

Exclusion Criteria:

* Congenital malformation neurological, cardiac, respiratory, vascular and cutaneous.
* A proven episode of materno-fetal infection

Ages: 27 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn of corrected age between 27 SA and 42 SA with at least 72 hours of postnatal age
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-03-24 (Estimated); Study Completion 2018-03-24 (Estimated)

PRIMARY OUTCOMES:
Measurement of the mean value of the perfusion index (PI) measured on the right hand | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France